CLINICAL TRIAL: NCT02295631
Title: A Comparison of Conventional Tube and ETView VivaSight SL Tube for Tracheal Intubation in Patients With a Cervical Spine Immobilisation. A Randomized Cross-over Manikin Trial.
Brief Title: ETI During Spinal Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/42
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Intubation; Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETI during immobilized spine (oral intubation) (Experimental): intubation with immobilized cervical spine endotracheal intubation with immobilized cervical spine
  Interventions: Device: Standard tracheal tube; Device: ETView VivaSight SL
- ETI during immobilized spine (nasal intubation) (Experimental): intubation with immobilized cervical spine endotracheal intubation with immobilized cervical spine
  Interventions: Device: Standard tracheal tube; Device: ETView VivaSight SL

INTERVENTIONS:
Device: Standard tracheal tube — ETI with standard tracheal tube and Macintosh laryngoscope
Device: ETView VivaSight SL — ETI with ETView VivaSight SL

SUMMARY:
The aim of this study was to compare time, success rates of different tracheal tubes (standard tube and ETView VivaSight SL) for intubation with an immobilized cervical spine in a standardized manikin model.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medicine personnel (physicians, nurses, paramedics)

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of first, second and third intubation attempts and overall effectiveness of intubation by participants

SECONDARY OUTCOMES:
Intubation time | 1 day
  time in seconds required for a successful intubation attempt
Cormack-Lehane grading | 1 day
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading (grade 1-4)
Preferred ETI device | 1day
  participants were asked which method of ETI they would prefer in a real-life resuscitation.

CONTACTS AND LOCATIONS:
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland